CLINICAL TRIAL: NCT06433700
Title: Risk of Revision and Other Complications Following Knee Arthroplasty in Patients Previously Exposed to Bariatric Surgeries: A Nationwide, Register-based Study
Brief Title: Risk of Revision Following Knee Arthroplasty in Bariatric Surgery Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Saber Muthanna Saber, Principal Investigator, PhD Fellow, Bispebjerg Hospital
Other Study IDs: p-2023-14433
Record Dates: First submitted 2023-09-07; First posted 2024-05-30 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Arthritis Knee; Bariatric Surgery Candidate; Prosthesis Failure; Prosthesis Survival; Prosthesis-Related Infections
Keywords: arthroplasty; revision; bariatric
MeSH Terms: conditions — Prosthesis Failure; Prosthesis-Related Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BAS group: Patients who received bariatric surgery prior to their knee arthroplasty
  Interventions: Other: BAS
- Non-BAS group: Patients who did not receive bariatric surgery prior to their knee arthroplasty
  Interventions: Other: Non-BAS

INTERVENTIONS:
Other: BAS — NOMESCO (Nordic Medico-Statistical Committee) Classification of Surgical Procedures (KJDF10 & KJDF11 [gastric bypass]; KJDF20 & KJDF21 [gastric banding]; KJDF40, KJDF41, KJDF96 & KJDF97 [gastric sleeve]).
  Groups: BAS group
Other: Non-BAS — Patients without BAS codes
  Groups: Non-BAS group

SUMMARY:
Previous studies have investigated the outcomes of Knee Arthroplasty (KA) following Bariatric Surgery (BAS), but with substantial limitations as not stratifying for Body Mass Index (BMI) at time of KA or not addressing the type of BAS (gastric bypass, banding or sleeve). Since BMI varies greatly in patients with previous BAS, it is likely that BMI affects outcomes after KA in BAS-operated patients.

The investigators believe that stratifying for BMI would explain the contradictions with the previous research in this patient group when it comes to the risk of revision after KA.

ELIGIBILITY:
Inclusion Criteria:

* Primary knee arthroplasty due to osteoarthritis

Exclusion Criteria:

* Primary knee arthroplasty due to traumatic osteoarthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will include patients with primary/idiopathic or secondary (due to meniscus or cruciate ligament lesion) osteoarthritis (OA) who received primary KA in the period from 2011 and 2 years earlier to data-extraction date. Patients will be identified from the DKR. Patients are followed for 2 years, until first revision, death or migration, whichever comes first.
Sampling Method: Probability Sample
Enrollment: 90000 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Hazard rate of Revision due to any cause | within 90 days and within 2 years
  Revision surgery is defined as surgery with debridement and/or exchange of at least one component
Hazard rate of Revision due to infection | within 90 days and within 2 years
  Our definition of infection is adapted from the European Bone and Joint Infection Society (EBJIS) criteria as at least one of the following A. An indication of deep infection is reported to the Danish knee arthroplasty register (DKR) by the surgeon on revision surgery B. At least 2 deep-tissue samples of phenotypically indistinguishable bacteria isolated from at least 3 deep-tissue samples C. One or more positive intraoperative samples from a closed fluid aspirate AND a biopsy (fluid AND tissue) of phenotypically indistinguishable bacteria isolated.

SECONDARY OUTCOMES:
Hazard rate of Knee related antibiotic use within 30- and 90-days following KA | within 30- and 90-days following KA
  the use of one of the following oral antibiotics: dicloxacillin, flucloxacillin, phenoxymethylpenicillin, amoxicillin, oral ciprofloxacin, roxithromycin, linezolid, cefuroxime and cefalexin
Hazard rate of Antibiotic use due to other causes | within 30- and 90-days following KA
  the use of one of oral antibiotics other than those that were mentioned in outcome 3.
Mortality | 2 years postoperatively
  Mortality registered in the Danish Civil Registration System (DCRS) by date

CONTACTS AND LOCATIONS:
Overall Officials: Søren Overgaard, MD,DMSc,Prof, Study Director — Department of orthopedic surgery, Bispebjerg University Hospital, Denmark
Locations (1):
- Orthopaedic department, Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: SAP outlined (2024-05-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT06433700/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Detailed SAP (2024-11-26): https://cdn.clinicaltrials.gov/large-docs/00/NCT06433700/SAP_001.pdf